CLINICAL TRIAL: NCT04354558
Title: Epidemiology and Outcomes of Critically Ill Patients With Covid 19: a French Single Centre Experience
Brief Title: French Single Centre Experience of Critically Ill Patients With Covid 19
Acronym: CovidAmiens20
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2020_843_0026
Record Dates: First submitted 2020-04-06; First posted 2020-04-21 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Epidemiology; Sars-CoV2; COVID 19; Critical Care; Prognostic; Survival
Keywords: Epidemiology; Sars-CoV2; COVID 19; critical care; prognostic; survival
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — alveolar liquid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- survival patients: The cohort will be dichotomised in survival/non-survival groups according to the issue during ICU stay
- non-survival patients: The cohort will be dichotomised in survival/non-survival groups according to the issue during ICU stay

SUMMARY:
Since the outbreak of a syndrome of acute respiratory distress associated to a novel coronavirus 2 (SARS-Cov2) that began in China, Europe and France have to face a sanitary emergency with critically care support when the patient evolves to an acute respiratory distress (ARDS). In the context of supply shortages (ventilators, bed capacities) that countries have to deal with, data were lacking of characteristics and outcomes of patients admitted to intensive care unit (ICU). the purpose of this project is to report the epidemiology and the outcomes of a French cohort of critically ill patients with SARS-Cov2

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* patient with positive rRT PCR of SARS Cov2 on a sample of nasopharyngeal swab
* admission in intensive care unit

Exclusion Criteria:

* patient under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with SARS Cov2 admitted in ICU
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Variation of age between critically ill patients with SARS Cov2 admitted in ICU with non critically ill patients with SARS Cov2 admitted in ICU | from day 1 of admission
  Variation of age between critically ill patients with SARS Cov2 admitted in ICU with non critically ill patients with SARS Cov2 admitted in ICU
Variation of medical history between critically ill patients with SARS Cov2 admitted in ICU with non critically ill patients with SARS Cov2 admitted in ICU | from day 1 of admission
  Variation of medical history between critically ill patients with SARS Cov2 admitted in ICU with non critically ill patients with SARS Cov2 admitted in ICU
Variation of chronic drug used between critically ill patients with SARS Cov2 admitted in ICU with non critically ill patients with SARS Cov2 admitted in ICU | from day 1 of admission
  Variation of chronic drug used between critically ill patients with SARS Cov2 admitted in ICU with non critically ill patients with SARS Cov2 admitted in ICU
Variation of chest CT scan at admission, between critically ill patients with SARS Cov2 admitted in ICU with non critically ill patients with SARS Cov2 admitted in ICU | from day 1 of admission
  Variation of chest CT scan at admission, between critically ill patients with SARS Cov2 admitted in ICU with non critically ill patients with SARS Cov2 admitted in ICU
Variation of respiratory support at ICU admission, between critically ill patients with SARS Cov2 admitted in ICU with non critically ill patients with SARS Cov2 admitted in ICU | from day 1 of admission
  Variation of respiratory support at ICU admission, between critically ill patients with SARS Cov2 admitted in ICU with non critically ill patients with SARS Cov2 admitted in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Osama Abou Arab, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beyls C, Huette P, Viart C, Mestan B, Haye G, Guilbart M, Bernasinski M, Besserve P, Leviel F, Witte Pfister A, De Dominicis F, Jounieaux V, Berna P, Dupont H, Abou-Arab O, Mahjoub Y. Mortality of COVID-19 Patients Requiring Extracorporeal Membrane Oxygenation During the Three Epidemic Waves. ASAIO J. 2022 Dec 1;68(12):1434-1442. doi: 10.1097/MAT.0000000000001787. Epub 2022 Oct 2. PMID 36194473
- [Derived] Beyls C, Hermida A, Bohbot Y, Martin N, Viart C, Boisgard S, Daumin C, Huette P, Dupont H, Abou-Arab O, Mahjoub Y. Automated left atrial strain analysis for predicting atrial fibrillation in severe COVID-19 pneumonia: a prospective study. Ann Intensive Care. 2021 Dec 7;11(1):168. doi: 10.1186/s13613-021-00955-w. PMID 34874509